CLINICAL TRIAL: NCT03977948
Title: Qualitative and Systemic Assessment of a Family Health Nurse Intervention Through Play, Which Aims to Prepare an Inpatient Child and His or Her Parents for Heart Surgery
Brief Title: Qualitative and Systemic Assessment of a Nurse Intervention an Inpatient Child and His or Her Parents
Acronym: EVALINF
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01623-52
Record Dates: First submitted 2019-05-20; First posted 2019-06-06 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2019-05

CONDITIONS: Anxiety State; Surgery; Pediatric Disorder
Keywords: cardiac surgery pediatric; preoperative anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured systemic interview — Semi-structured systemic interviews will be conducted with families who have benefited from the preparation for surgery through play. Other tools such as the logbook and the socio-demographic questionnaire will also be used. The themes that will emerge from these interviews will provide a better understanding of what these families are going through, how the proposed intervention may or may not have met their expectations, and provide insights so that health care services can build their own surgical preparation programs.

SUMMARY:
The hospitalization of a child for cardiac surgery is a major event in a family's life. Some factors induced by surgery can have serious psychological consequences and cause high stress and anxiety in the child but also in the parents. Many interventions have been tested to reduce this anxiety generated by apprehension of the surgical procedure, but there is no evidence to date that would allow health care services to effectively prepare these families for surgery. The authors encourage researchers to continue research on this subject in order to confirm or refute their results.

DETAILED DESCRIPTION:
The hospitalization of a child for surgery is a major event that can disrupt a family's life. Indeed, whatever the degree of severity and type of pathology that leads to hospitalization, a stay in hospital is often synonymous with stress and fear, both for the child and for parents. A lack of knowledge of care procedures, the feeling of not being able to control the situation and a lack of explanations in terms adapted to their age are all factors that contribute to the vulnerability of children hospitalized for surgery.

Preoperative anxiety can be defined as an overflow of the child's ability to cope with stress, induced by the fear of surgery. Significant preoperative anxiety could increase the risk of post-operative complications and promote emotional and behavioural disorders such as: insecurity, guilt, anger, anger, regression, withdrawal or rebellion, it could also have the effect of limiting the child's ability to cope with surgery, encouraging negative behaviours related to health care, but also inhibiting post-operative recovery. These behavioural disorders induced by preoperative anxiety may persist once hospitalization is completed and the family returns home. In addition, if the operating experience is negative, the child may develop separation anxiety or even phobia following surgery and in extreme cases acute stress or even post-traumatic stress. The risk for the child to develop one of these disorders following surgery is increased by the frequency and duration of the anxiety episodes to which he or she will be subjected.

Parents of children hospitalized for surgery would also experience very high stress, related to their perception of their child's state of health, apprehension of invasive treatments, as well as fear of sequelae that could be caused by certain invasive treatments or because of their child's pathology. It is therefore important, during hospitalization and surgery, to take into consideration the anxiety of the child, but also of his or her parents, and to consider how best to manage this anxiety in order to prevent complications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years hospitalized for open-heart surgery
* Children who have participated in the daily surgical preparation activity provided by M3 nurses to families whose child is hospitalized for open-heart surgery.
* Ability to understand and speak French
* The parent (biological or adoptive) must have participated in the activity of preparation for surgery.

Exclusion Criteria:

* Child with a psychological pathology diagnosed in the medical file or notified by the parents at the first contact (autism, depression...)
* Children with cognitive problems that do not allow the interviews diagnosed in the medical file or notified by the parents at the first contact to take place
* Genetic syndrome

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: The child with his family
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 1 day
  parents's and children's feelings about the nurse's preparation : Advantages and disadvantages, open- Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No